CLINICAL TRIAL: NCT00300040
Title: Phase II, Multi-Center,Single-Blind,Placebo-Controlled Study,Evaluating Safety & Feasibility of HBOC-201 (Wound Healing Patients With Peripheral Vascular Disease & Undergoing Lower Limb Amputation Due to Critical Lower Limb Ischemia
Brief Title: Safety/Feasibility Study of HBOC-201 in Amputation at/Below Knee From Critical Lower Limb Ischemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Very slow enrollment.Study entry criteria not in line w/local standards of care
Sponsor: Biopure Corporation (Industry)
Responsible Party: Biopure, Biopure
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIOSA001/BIOEU001
Record Dates: First submitted 2006-03-06; First posted 2006-03-08 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Peripheral Vascular Disease
Keywords: Amputation; Lower limb; Critical Limb Ischemia; residual limb; Peripheral Vascular Disease; re-amputation; Lower Limb Ischemia; PVD
MeSH Terms: conditions — Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia | interventions — HBOC 201; Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Hemoglobin glutamer 250 - bovine
  Interventions: Drug: Hemoglobin glutamer 250 - bovine
- 2 (Active Comparator): 6% Hydroxyethylstarch
  Interventions: Drug: 6% Hydroxyethylstarch

INTERVENTIONS:
Drug: Hemoglobin glutamer 250 - bovine — intravenous - 250ml/dose - 32.5g Hb (Concentration 13 +/- 1g/dL)
  Other Names: Hemopure; HBOC-201
  Arms: 1
Drug: 6% Hydroxyethylstarch — 250ml for intravenous infusion
  Other Names: HAES-steril®
  Arms: 2

SUMMARY:
The purpose of this study is to assess the safety and feasibility of HBOC-201 in increasing adequate wound healing in patients with severe peripheral vascular disease who are undergoing lower limb amputation.

The hypothesis is that HBOC-201 will pass through the partially occluded lesions in the peripheral arteries in the lower extremity and promote the wound healing process by delivering oxygen to the oxygen deprived tissues. This will reduce the incidence of lower limb wound complications at 60 days post-surgery and may reduce the incidence of a second amputation.

DETAILED DESCRIPTION:
This is a Phase II, single-blinded, prospectively randomized, parallel-group, placebo controlled study that will evaluate the safety and feasibility of HBOC-201 when administered therapeutically to patients with a peripheral vascular occlusive disorder and who are undergoing lower limb amputation due to critical lower limb ischemia. Subjects will be randomized (1:1) to receive either HBOC-201 or a colloid control (HAES-steril® 6%).

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 ≤ 75 years of age
* Scheduled amputation at or above ankle joint, or a more proximal location but below or through the knee joint
* Documented severe lower extremity peripheral artery occlusive disease confirmed by clinical symptoms of critical limb ischemia and:

  * Frankly gangrenous tissue that merits amputation or
  * Angiographic evidence of occlusive peripheral artery disease within one month of screening
* Participant or legal representative signs informed consent
* Willingness to follow study instructions and follow-up visits

Exclusion Criteria:

* No informed consent is obtained
* If medically inappropriate to administer 250 mL colloidal solution daily for 4 consecutive days
* Uncontrolled hypertension (BP > 160/90 mm Hg) despite 2 antihypertensive meds or BP > 180/100 mm Hg if untreated
* Severe liver dysfunction defined by Total Bilirubin > 3 mg/dL or twice the normal limit of serum AST or ALT
* Symptomatic CVD diagnosed w/ in last 6 months or known high grade carotid stenosis
* Any severe or unstable medical condition that might interfere w/ the evaluation of study medication
* Cardiogenic shock (cardiac index < 2 L/min/m2, PCWP > 18 mm Hg)
* Amputation above knee joint or below ankle joint
* Any amputation whereby primary skin closure not technically feasible
* Candidate for percutaneous or surgical revascularization
* Cardiac failure defined by a NY class III/IV or left ventricular ejection fraction < 30%
* Life expectancy < 60 days
* Systemic mastocytosis
* Previously demonstrated beef product allergy
* Myocardial infarction w/ in 30 days
* Participation in another trial w/ in last 30 days
* Woman who is pregnant or breastfeeding
* Amputation with known infection at site of skin closure
* Renal dysfunction requiring dialysis, or serum creatinine level 2.5 mg/dL
* Peripheral vascular occlusion from cardio arterial emboli
* Uncontrolled diabetes blood glucose ≥ 400 mg/dL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-05; Primary Completion 2008-06 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Mortality at 60 days post amputation procedure | 60(±7 days) post-procedure follow-up visit

SECONDARY OUTCOMES:
30 day follow up mortality; Complete wound healing 30, 60 day follow up; Time to complete wound healing; Re-amputation 60 days; Hospital, ICU & rehab days; TcPO2 change; Quality of Life; Delayed wound healing/complications; Rehospitalization; Surgeries | 15(±3 days) , 30(±7 days) and 60(±7 days) post-procedure follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: A. Gerson Greenburg, MD, Ph.D., Study Director — Biopure Corporation
Locations (5):
- South Africa (4):
  - Johannesburg Hospital, Johannesburg, Guateng
  - Milpark Hospital, Parktown West, Guateng
  - Pretoria Academic Hospital, Pretoria, Guateng
  - University of Stellenbosch, Tygerburg
- John Radcliffe Hospital, Headington, Oxfordshire, United Kingdom